CLINICAL TRIAL: NCT02754037
Title: Non-alcoholic Fatty Liver Disease Parametric PET (FLiPP) Study
Acronym: FLiPP
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 840422; R01DK124803-01A1 (NIH)
Record Dates: First submitted 2016-04-26; First posted 2016-04-28 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD); Non-alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood plasma/serum will be banked at the University of California, Davis GI Biobank for future liver-related study use in -80°C freezer. Samples will be used for liver related studies. Potential future analyses of plasma samples could include fatty liver metabolomics analyses. All future Sample specimens will be stored for as long as they are viable (for up to 20 years). Dr. Medici and her study staff will maintain records of the storage location and have access to them.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Fluorodeoxyglucose (FDG) positron emission tomography (PET) — This imaging method uses radiotracers for functional analysis of liver inflammation. It does involve placement of an intravenous catheter and a radiotracer. One blood sample (10cc) will be drawn after PET scan using a butterfly method with the time recorded. The blood sample will be centrifuged in the Main Hospital to get the plasma and a well counter will be used to calculate the radioactivity in the plasma as per established protocol. Potential risks from an intravenous catheter insertion and blood draw include pain, minimal blood loss and local erythema. Radiotracer exposure from FDG-PET is minimal and has been well-characterized. Radiation Use Committee approval has been obtained for FDG-PET use.
Other: Magnetic resonance imaging (MRI) — Novel non-invasive MRI based tools to assess liver fat and fibrosis. Potential risks include a sensation of claustrophobia. No contrast dye is used and thus no risk of contrast allergy. Inflammation of the liver may be assessed by MRI software after processing of images and does not require additional patient involvement or change in MRI protocol.
  Other Names: Magnetic resonance proton density fat fraction (MR-PDFF), Magnetic resonance elastography (MRE)
Radiation: PET Explorer — Similar to the regular PET-Scan, this imaging method uses radiotracers to scan multiple organs of the body. It does involve placement of an intravenous catheter and a radiotracer. One blood sample (10cc) will be drawn after PET scan using a butterfly method with the time recorded. The blood sample will be centrifuged in the Main Hospital to get the plasma and a well counter will be used to calculate the radioactivity in the plasma as per established protocol. Potential risks from an intravenous catheter insertion and blood draw include pain, minimal blood loss and local erythema. Radiotracer exposure from FDG-PET is minimal and has been well-characterized. Radiation Use Committee approval has been obtained for FDG-PET use.

SUMMARY:
The goal of this study is to evaluate non-invasive imaging techniques for determining liver steatosis (fat), inflammation (abnormal tissue swelling), and fibrosis (abnormal tissue scarring).In addition, the study group will be using other test measures including personal demographics, laboratory blood test results, and imaging measurements to determine the severity of NAFLD (non-alcoholic fatty liver disease), NASH (non-alcoholic steatohepatitis), inflammation, and fibrosis.

DETAILED DESCRIPTION:
The study group proposes to evaluate the role of fluorodeoxyglucose (FDG) positron emission tomography (PET) in the determination of steatohepatitis and in combination with MRI for detection, differentiation and quantitation of liver steatosis, steatohepatitis and fibrosis in correlation to liver biopsy. Patient enrolled in this will already have had their liver biopsy or will be undergoing liver biopsy as a part of their clinical care as determined by their provider and will not be getting biopsies solely to be enrolled in the study. Current treatment options for patients that liver biopsy is being performed are limited to lifestyle changes and vitamin E for patients without diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >18 years age
2. Patients who had or will have a liver biopsy as standard of care for fatty liver disease and have risk factors for NASH. Liver biopsy needs to be within 6 months of planned imaging.
3. Patients undergoing bariatric surgery and will have a liver biopsy as standard of care.
4. Ability to provide informed consent.

Exclusion Criteria:

1. History of alcohol abuse, chronic hepatitis B or C, or other chronic liver disease other than non-alcoholic fatty liver disease.
2. Pregnant women
3. Prisoners
4. Claustrophobic to MRI
5. Allergic to FDG dye
6. Patients who are unable to lie in the scanner for one hour

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes those who are scheduled to have bariatric surgery (weight loss surgery) or have had a liver biopsy within the past six months with a diagnosis of Non-Alcoholic Fatty Liver Disease (NAFLD) or Non-Alcoholic Steatohepatitis (NASH). These
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-04-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
PET scan parameters correlated with biopsy findings | one year
  PET scan parameters correlated with biopsy findings (NAFLD Activity Score as per NASH-CRN)

CONTACTS AND LOCATIONS:
Overall Officials: Guobao Wang, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared

REFERENCES:
- [Derived] Sarkar S, Chen S, Spencer B, Situ X, Afkarian M, Matsukuma K, Corwin MT, Wang G. Non-Alcoholic Steatohepatitis Severity Associates with FGF21 Level and Kidney Glucose Uptake. Metab Syndr Relat Disord. 2021 Nov;19(9):491-497. doi: 10.1089/met.2021.0055. Epub 2021 Aug 26. PMID 34448598
- See also: Learn more or sign up for the study here! — https://studypages.com/s/non-invasive-evaluation-of-liver-steatosis-inflammation-and-fibrosis-780989/